CLINICAL TRIAL: NCT02010489
Title: The Impact of a Pre-Operative Exercise Program on Fitness Outcomes Following Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H2013:388
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Obesity
Keywords: Bariatric Surgery; Exercise; Physical Fitness
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Following randomization, the control group will receive usual preoperative care consisting of two to four multidisciplinary visits over six months. During this time, patients will be provided with exercise counseling through the team kinesiologist. They will complete a behavior modification program called Craving ChangeTM and must achieve usual goals of lifestyle and dietary modification, along with modest weight loss of approximately 5%, in order to be scheduled for surgery. Patients will also complete a liquid diet consisting of 900 calories per day for two weeks prior to their procedure in order to reduce intra-abdominal obesity and facilitate the procedure.
- 12 Week Exercise Program (Other): The intervention group will undergo standard pre-operative care and will also be enrolled in a 12-week exercise program at the Reh-Fit Centre in Winnipeg. The Reh-Fit Centre is a non-profit organization with the mission to enhance the health and wellbeing of its members and the community by providing innovative health and fitness services. The intervention will be offered at no cost to the patient. It will involve regular supervised exercise sessions at the Reh-fit centre three times per week. Most patients will complete the intervention prior to commencing the liquid diet but will otherwise discontinue the program while on the diet two weeks prior to surgery.
  Interventions: Other: 12 week Exercise Program

INTERVENTIONS:
Other: 12 week Exercise Program — Patients will be provided with a tour of the Reh-Fit Centre, exercise prescription, and supervised exercise session. The exercise prescription consists of 3 weekly 60-minute sessions, each with 10 minutes warm-up, 30 minutes endurance, 20 minutes strength training and 5 minutes cool-down. The program is overseen by an accredited Exercise Physiologist. Initial exercise intensity is determined by the kinesiologist and based on the patient's baseline fitness level. Goal intensity of endurance activity is based on the heart rate reserve (HRR) method. This is captured with a heart rate monitor at initial assessment and recorded on exercise logs. There are check-ins at each exercise session to determine progress (time, reps, weight, sets, etc). Endurance activities include treadmill, elliptical, walking, and aerobics. Strength training includes upper body, lower body, and trunk circuits. Patients will be asked to attend three weekly sessions at the Reh-Fit Centre.
  Arms: 12 Week Exercise Program

SUMMARY:
BACKGROUND: Obesity is a global epidemic and Canada has one of the highest obesity rates in westernized countries. Obesity has many health related complications, including high blood pressure, high cholesterol, diabetes, sleep apnea and osteoarthritis. Bariatric surgery is the most effective way of achieving long-term weight loss and treating the complications of obesity. There is good evidence to support the relationship between physical activity and weight loss following bariatric surgery. While the period leading up to surgery is considered an important opportunity for lifestyle modification, evidence to support recommendations for a supervised preoperative exercise intervention is lacking.

OBJECTIVES: The objective of this study is to measure the short and intermediate-term benefits of a preoperative exercise intervention on patients awaiting publicly funded bariatric surgery in Manitoba. The primary outcome will be improvement in general exercise capacity as measured by change in 6-minute walk test (how far a person can walk on a flat surface in 6 minutes). Other outcomes will include excess weight loss, change in body composition, strength testing and irisin bloodwork & muscle biopsy.

HYPOTHESIS: It is hypothesized that preoperative exercise will result in improved exercise capacity and general fitness in the short and intermediate-term post-bariatric surgery.

METHODS: Patients who are awaiting publicly funded bariatric surgery in Manitoba will be offered the opportunity to participate in a randomized study between usual preoperative care (n=35) and usual care plus a supervised exercise program (n=35). Usual care will involve multidisciplinary evaluation and preoperative counseling with a kinesiologist. In the intervention group, patients will participate in a 12-week supervised exercise program at the Reh-fit Centre.

RESULTS: The study will determine the short and intermediate-term benefits of a preoperative exercise intervention on general fitness and exercise capacity as well as weight loss post-bariatric surgery. It is an important opportunity for collaboration between a multidisciplinary health care team and a medically-certified community fitness centre. Currently there are approximately 200 patients undergoing public bariatric surgery annually in Manitoba. If this study demonstrates a benefit to preoperative exercise, the results will be used to support an application to Manitoba Health for routine implementation of a similar intervention for all patients awaiting publicly funded bariatric surgery. It will also be used to support an application for a larger multi-institutional study of preoperative exercise at several Canadian bariatric centres.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 years or older
* Awaiting publicly funded bariatric surgery through the Centre for Metabolic and Bariatric Surgery
* Must be undergoing surgery within six months of tentative approval (usual timeline)
* Must be able to participate in an exercise program at the Reh-Fit Centre in Winnipeg. There will be a home option for some of the activities but patients will be expected to attend at least one of three sessions at the Reh-Fit Centre weekly

Exclusion Criteria:

* Orthopedic, neurologic or cardiopulmonary conditions that preclude moderately strenuous exercise
* In general, patients are not considered candidates for bariatric surgery if they are wheelchair bound or cannot tolerate moderate physical activity.
* Patients will also be excluded if they are unable to commit to attending regular sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test (6MWT) | Pre-Intervention
  The 6MWT is a validated measure of physical fitness (22) and involves measuring the distance a patient walks unassisted in six minutes at a self-selected pace.
6 Minute Walk Test | Post Intervention (12 weeks)
6 Minute Walk Test | Post Operative (3 months)
6 Minute Walk Test | Post Operative (6 months)

SECONDARY OUTCOMES:
Anthropometric Measurements | Pre-Intervention
  Includes:
  1. Height (SECA 242 Electronic stadiometer)
  2. Weight (SECA 645 Multifunctional handrail scale)
  3. BMI (kg/m2)
  4. Neck circumference
  5. Waist and hip circumference
Anthropometric Measurements | Post Intervention (12 weeks)
  Includes:
  1. Height (SECA 242 Electronic stadiometer)
  2. Weight (SECA 645 Multifunctional handrail scale)
  3. BMI (kg/m2)
  4. Neck circumference
  5. Waist and hip circumference
Anthropometric Measurements | Post Operative (3 months)
  Includes:
  1. Height (SECA 242 Electronic stadiometer)
  2. Weight (SECA 645 Multifunctional handrail scale)
  3. BMI (kg/m2)
  4. Neck circumference
  5. Waist and hip circumference
Anthropometric Measurements | Post Operative (6 months)
  Includes:
  1. Height (SECA 242 Electronic stadiometer)
  2. Weight (SECA 645 Multifunctional handrail scale)
  3. BMI (kg/m2)
  4. Neck circumference
  5. Waist and hip circumference
Body Composition | Pre-Intervention
  Measured using Dual-energy X-ray Absorptiometry
Body Composition | Post Operative (6 months)
  Measured using Dual-energy X-ray Absorptiometry
Strength Measures | Pre-Intervention
  Includes
  1. Chair to stand test
  2. Half squat test
  3. Hand grip test
Strength Measures | Post Intervention (12 weeks)
  Includes
  1. Chair to stand test
  2. Half squat test
  3. Hand grip test
Strength Measures | Post Operative (3 months)
  Includes
  1. Chair to stand test
  2. Half squat test
  3. Hand grip test
Strength Measures | Post Operative (6 months)
  Includes
  1. Chair to stand test
  2. Half squat test
  3. Hand grip test
Other Measures | Pre-Intervention
  Includes:
  1. Accelerometer Physical Activity Level (Actigraph: Pensacola, FL)
  2. Laval Health Related Quality of Life Questionnaire
  3. Satisfaction Survey
Other Measures | Post Intervention (12 weeks)
  Includes:
  1. Accelerometer Physical Activity Level (Actigraph: Pensacola, FL)
  2. Laval Health Related Quality of Life Questionnaire
  3. Satisfaction Survey
Other Measures | Post Operative (3 months)
  Includes:
  1. Accelerometer Physical Activity Level (Actigraph: Pensacola, FL)
  2. Laval Health Related Quality of Life Questionnaire
  3. Satisfaction Survey
Other Measures | Post Operative (6 months)
  Includes:
  1. Accelerometer Physical Activity Level (Actigraph: Pensacola, FL)
  2. Laval Health Related Quality of Life Questionnaire
  3. Satisfaction Survey
Physical Activity Level | Pre-Intervention
  Measured using accelerometers
Physical Activity Level | Mid Intervention (6 weeks)
  Measured using accelerometers
Physical Activity Level | Post Operative (6 months)
  Measured using accelerometers
Irisin bloodwork | At study enrollment/pre-intervention
  Irisin is a recently discovered peptide secreted by the skeletal muscle. It has been proposed that this novel peptide is secreted by muscle in response to exercise training and trigger cross talk between skeletal muscle and other organs. In fact, the beneficial effects of irisin would be elicited through an up-regulation of energy consumption within adipocytes, which results in glucose tolerance improvement and increase in endurance performance. Until now, one study investigated the predictor of changes in irisin following a bariatric surgery. However, no study has yet investigated whether a pre-surgery physical activity program contributes to the change in irisin level in severely obese patients.
Irisin bloodwork | Post intervention/Pre-Surgery
Irisin Bloodwork | Post operative (while in hospital)
Irisin Bloodwork | Post operative (3 months)
Irisin Bloodwork | Post Operative (6 months)
Muscle Biopsy (optional) | Intra operative

CONTACTS AND LOCATIONS:
Overall Officials: Krista Hardy, MD, Principal Investigator — Assistant Professor, University of Manitoba
Locations (1):
- Centre for Metabolic and Bariatric Surgery, Victoria General Hospital, Winnipeg, Manitoba, Canada